CLINICAL TRIAL: NCT03988361
Title: Evaluation of Embryo Quality After Enrichment of Non-apoptotic Spermatozoa Using Magnetic-activated Cell Sorting (MACS): Study on Sibling Oocytes.
Brief Title: Selection of Non Apoptotic Human Sperm for in Vitro Fertilization by Using Magnetic Activated Cell Sorting (MACS)
Acronym: MACS-HS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Ileana Mateizel, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: 2018-183
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Half of the mature oocytes of the same patient will be injected with sperm obtained after DGC only (conventionally semen preparation).
- Study group: Half of the mature oocytes of the same patient will be injected with sperm obtained after DGC and MACS.
  The sperm used in this group is considered to be enriched in non apoptotic cells.
  Interventions: Diagnostic Test: Magnetic Activated Cell Sorting

INTERVENTIONS:
Diagnostic Test: Magnetic Activated Cell Sorting — At the moment of ICSI, sibling mature oocytes will be inseminated with spermatozoa from Study group or from Control group. Following ICSI, all the inseminated oocytes will be individually cultured in the same conditions in the same culture dish. The choice of embryo(s) for transfer will be based on embryo quality. The supernumerary good-quality embryos from both arms will be frozen for further use.
  Groups: Study group

SUMMARY:
This clinical study has been organised to help improve the embryo quality in couples having high rate of sperm showing apoptotic signs. For this, the investigators intend to use a procedure (MACS: magnetic-activated cell sorting) that allows the identification and the removal of the apoptotic sperm cells. This procedure will increase the chance of using non-apoptotic sperm during in vitro fertilization via Intracytoplasmic Sperm Injection (ICSI). By using this procedure the investigators aim to increase the rate of embryos with good quality for these particular couples.

DETAILED DESCRIPTION:
Studies of infertile couples have demonstrated that male factor plays a role in infertility. Spermatozoa can present damages at molecular levels that have an effect on fertilization and embryo development. One of these molecular damages is represented by DeoxyriboNucleic Acid (DNA) fragmentation whose negative impact on embryological outcome appears during genome activation after fertilization and is also correlated with increased miscarriage rate.

DNA fragmentation represents one of the late manifestations of apoptosis. Identification of spermatozoa showing DNA fragmentation (apoptotic spermatozoa) requires fixation and staining. Therefore this method cannot be applied in clinical practice to select for non-apoptotic spermatozoa for ICSI. However, this selection is possible by using magnetic-activated cell sorting (MACS). The procedure is based on the identification and depletion of spermatozoa showing the early marker of apoptosis, namely the externalization of phosphatidylserine (PS), by using the ability of Annexin V to recognize this antigen in the plasma membrane of apoptotic sperm cells. After MACS, the fraction that is enriched in non-apoptotic cells (Annexin V-negative cells) can be further used for clinical application.

The MACS system makes use of a separation column placed in a magnetic field, and of Annexin-V reagent labeled with paramagnetic beads.

Initially, the semen sample will be subject to Density Gradient Centrifugation (DGC). The sample obtained will be divided in 2 fractions: one fraction will be subject to magnetic sorting (fraction 1) and the other fraction will represent the control (no sorting; fraction 2).

The cells from fraction 1 will be incubated with Annexin-V and then passed through the separation column located in a magnetic field. The apoptotic cells (Annexin V-positive cells) will be selectively retained in the column. The non-apoptotic cells, not being labeled by Annexin V, will pass through the column and will be collected for further use.

At the moment of ICSI, sibling mature oocytes will be inseminated with spermatozoa from fraction 1 (enriched in non-apoptotic cells) or from fraction 2 (control, conventionally prepared spermatozoa). Following ICSI, all the inseminated oocytes will be individually cultured in the same conditions in the same culture dish. The choice of embryo(s) for transfer will be based on embryo quality. The supernumerary good-quality embryos from both arms will be frozen for further use.

The present study aims to determine whether the use of MACS improves the embryo quality/utilization rate in couples with high sperm DNA fragmentation rate. To avoid inter-patient variation, the study is design as a sibling oocyte study. Descriptive statistics will be performed by analysing median, mean, proportions, standard deviation, ranges and 95% confidence intervals as appropriate. Standard parametric and non-parametric tests will be used, as appropriate, to compare primary and secondary outcomes between groups. Sample size calculation: a number of 142 mature oocytes in each arm will be necessary to achieve 80% power of detecting, as significant at the 5% level, an increase in the primary outcome measure from 13% in the control group to 26% in the experimental group.

ELIGIBILITY:
10.2 Inclusion Criteria

* Patients with poor embryo quality in the previous cycles:

  * Cycles with no embryo transfer due to insufficient embryo quality
  * "Freeze all" cycles without cryopreservation
  * Cycles with transfer of embryos with fair and/or poor quality
* Previous diagnostic semen analysis with minimum 30% DNA fragmentation
* ICSI cycles with fresh ejaculated semen with ≥1 mil spermatozoa after DGC.
* Minimum 6 mature oocytes after oocyte pick up.

10.3 Exclusion Criteria

* Cycles with frozen semen sample
* Cycles with testicular sample
* In vitro fertilization (IVF) cycles
* Cycles with pre-implantation genetic diagnosis
* In vitro maturation cycles

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples with poor embryo quality in the previous cycle at Centre of reproductive Medicine -Universitair Ziekenhuis Brussel and minimum 30% DNA fragmentation in the previous diagnostic semen analysis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
utilization rate | 2 years
  number of transferred and cryopreserved embryos per mature oocytes

SECONDARY OUTCOMES:
fertilization rate | 2 years
  number of fertilized oocytes per number of injected oocytes

IPD SHARING:
Plan to Share IPD: No